CLINICAL TRIAL: NCT01445860
Title: A Phase 1, Open-Label, Fixed-Sequence Study To Estimate The Effect Of Repeated Dosing Of PF-03882845 On The Pharmacokinetics Of A Single Dose Of Simvastatin In Healthy Adult Subjects
Brief Title: Drug-Drug Interaction Study Of Effect Of PF-03882845 On Simvastatin Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B0171013
Record Dates: First submitted 2011-07-11; First posted 2011-10-04 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: Human Volunteers
Keywords: DDI; pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Simvastatin/PF-03882845

INTERVENTIONS:
Drug: Simvastatin/PF-03882845 — Single dose 20 mg simvastatin on Day 1, 30 mg PF-03882845 once daily from Days 2 to 13, the single dose 20 mg simvastatin on Day 12.

SUMMARY:
The purpose of this study is to estimate the effect of multiple oral doses of PF-03882845 on the pharmacokinetics of simvastatin and simvastatin acid in healthy, adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and/or females of non-childbearing potential between the ages of 18 (or 21 based on country-specific age of consent) and 60 years, inclusive, at Screening. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical/safety laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2 inclusive; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Use of CYP3A4 inhibitors (eg, ketoconazole, ciprofloxacin, diltiazem) or inducers (eg, pheytoin, carbamazepine) or substrate (eg, simvastatin, quinidine) within 28 days or 5 half-lives (whichever is longer) prior to Day 1.
* Known history of hypersensitivity, allergy, severe adverse drug reaction or intolerance to simvastatin or other statins.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Composite (or Profile) of Pharmacokinetics | 15 days
  AUCinf, AUClast, Cmax, Tmax, t1/2 of simvastatin and simvastatin acid

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0171013&StudyName=Drug-Drug%20Interaction%20Study%20Of%20Effect%20Of%20PF-03882845%20On%20Simvastatin%20Pharmacokinetics